CLINICAL TRIAL: NCT01001117
Title: A Prospective Single-Center Clinical Trial to Evaluate the Feasibility of Laser Treatment of the Crystalline Lens in Subjects Having Elected to Undergo Lens Extraction and Intraocular Lens Implantation
Brief Title: Laser Treatment of the Crystalline Lens
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LensAR Incorporated (Industry)
Responsible Party: Director, Clinical & Regulatory Affairs, LensAR Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 52-00001-0000
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Cataract
Keywords: Cataract; Capsulotomy; Capsulorrhexis; Phacoemulsification
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser treated (Experimental): Eye treated with LensAR Laser System
  Interventions: Device: LensAR laser surgery
- Control Eye (Active Comparator): Contralateral eye treated with conventional phaco-emulsification
  Interventions: Device: Phaco-emulsification cataract surgery

INTERVENTIONS:
Device: LensAR laser surgery — Use of laser for cataract surgery
  Other Names: LensAR Laser System
  Arms: Laser treated
Device: Phaco-emulsification cataract surgery — Phaco-emulsification cataract surgery
  Other Names: Exact equipment varies
  Arms: Control Eye

SUMMARY:
The use of a femtosecond laser in cataract surgery that gives equivalent or improved results comapred to conventional phaco-emulsification surgery.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the feasibility of the LensAR laser system to surgically intervene within the crystalline lens. The primary goal of this initial study is to establish safety parameters as compared with conventional phacoemulsification procedures, and to evaluate the ability to provide an accurate and consistent anterior capsular opening (capsulotomy).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign and be given a copy of the written informed consent form.
* Subjects must have elected to undergo lens extraction and foldable monofocal IOL implantation (ideally of the same type), and then elect to have the LensAR laser surgery.
* Subjects must be willing and able to return for scheduled follow-up examinations for a minimum of 12 months after surgery.
* Central 8 mm of clear cornea without vascularization.

Exclusion Criteria:

* Subjects with prior anterior segment or vitreo-retinal surgical intervention in the eye to be treated.
* Subjects with lenticular cataracts with nuclear grading greater than Grade 4 on the LOCS III scale.
* Subjects who cannot attain ocular dilation of 7.0 mm.
* Subjects with anterior segment pathology in the eye to be treated that is not directly improved by lens extraction and IOL implantation.
* Subjects with residual, recurrent, active ocular or uncontrolled eyelid disease or any corneal abnormalities (including endothelial dystrophy, guttata, recurrent corneal erosion, etc.) in the eye to be treated.
* Subjects with ophthalmoscopic signs of keratoconus (or keratoconus suspect) in the eye to be treated.
* Subjects with a history of severe dry eye not responding to therapy.
* Subjects with macular degeneration, history of retinal detachment, or any other fundus findings that would pose a risk to safety or an acceptable visual outcome in the eye to be treated.
* Subjects with a history of herpes zoster or herpes simplex keratitis.
* Subjects who have a history of steroid-responsive rise in intraocular pressure, glaucoma, or are a glaucoma suspect.
* Subjects with diabetic retinopathy, autoimmune disease, connective tissue disease, pseudoexfoliation syndrome, or clinically significant atopic syndrome.
* Subjects on chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing, and any immuno-compromised subjects.
* Subjects who are using ophthalmic medication(s) other than artificial tears for treatment of ocular pathology including ocular allergy.
* Subjects using systemic medications with significant ocular side effects.
* Subjects who are pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.
* Subjects with known sensitivity to planned study concomitant medications.
* Subjects who are participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Capsulotomy a. Ease of opening b. Achievement of intended shape and size | Time of Surgery
Lens removal a. Ease of irrigation / aspiration (time) b. Reduced ultrasound phacoemulsification | Time of surgery
Posterior capsule rupture < 10% occurrence rate | Time of Surgery
Less than 5% of eyes should lose more than two lines of BSCVA | 3 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Naranjo, MD, Principal Investigator — Asociacion Para Evitar La Ceguera en Mexico IAP; Jorge VIllar, MD, Principal Investigator — Asociacion Para Evitar La Ceguera en Mexico IAP
Locations (1):
- Asociacion Para Evitar La Cuguera en Mexico IAP, Mexico City, Mexico

REFERENCES:
- [Derived] Tackman RN, Kuri JV, Nichamin LD, Edwards K. Anterior capsulotomy with an ultrashort-pulse laser. J Cataract Refract Surg. 2011 May;37(5):819-24. doi: 10.1016/j.jcrs.2010.11.030. Epub 2011 Mar 11. PMID 21397456